CLINICAL TRIAL: NCT06617793
Title: An Open-label, Multi-center, Phase 1/2 Study to Assess Safety, Efficacy, and Cellular Kinetics of YTB323 in Participants With Relapsing Multiple Sclerosis With Breakthrough Disease Activity During Previous Treatment With a Highly Efficacious Therapy
Brief Title: An Open-label Study to Assess the Safety, Efficacy, and Cellular Kinetics of YTB323 in Relapsing Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323N12101; 2024-512714-18 (Other: EU CTIS)
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Chimeric Antigen Receptor T cells; CAR-T; YTB323; Multiple Sclerosis; MS; Relapsing Multiple Sclerosis; RMS; breakthrough disease activity during previous treatment with a highly efficacious therapy; BD-HET
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YTB323 Cohort 1 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)
- YTB323 Cohort 2 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)
- YTB323 Cohort 3 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)
- YTB323 Cohort 4 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)

INTERVENTIONS:
Biological: rapcabtagene autoleucel (YTB323) — CAR-T cell suspension for intravenous infusion

SUMMARY:
This is an open-label, multi-center, non-confirmatory study to assess the safety, efficacy, and cellular kinetics of YTB323 in approximately 28 participants with Relapsing Multiple Sclerosis (RMS) with breakthrough disease activity during previous treatment with a highly efficacious therapy (BD-HET). The study design utilizes an ascending single dose design consisting of 3 sentinel cohorts followed by an expansion cohort.

DETAILED DESCRIPTION:
All participants in this study will receive YTB323. Both the participant and the study doctor will know the participant is getting YTB323. Participants will be given one dose of YTB323. Different groups of participants may receive a higher dose of YTB323, if proven to be safe for every participant at the lower dose. Participants are in this study for 2 years and will be followed for an additional 13 years in a long-term follow up study. The main question this trial is designed to answer: Is YTB323 treatment safe for participants with relapsing MS?

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, and able to communicate well with the investigator and comply with the requirements of the study
* Adequate renal, hepatic, cardiac, hematological, and pulmonary function
* Male or female participants, ≥18 years to ≤60 years at screening, with diagnosis of RMS according to the 2017 McDonald diagnostic criteria Evidence of recent (i.e. within 1 year) breakthrough disease activity while at least 6 months on a highly efficacious therapy (any of the following): rituximab (Rituxan®), ocrelizumab (Ocrevus®), natalizumab (Tysabri®), ofatumumab (Kesimpta®), ublituximab (Briumvi®) or evidence of breakthrough disease activity within 2 years after the latest alemtuzumab infusion (Lemtrada®).

Evidence of breakthrough disease activity is defined as one or more of the following:

1. Confirmed Clinical MS relapse
2. Persistent radiological activity defined by one of the following:

   * ≥2 T1 gadolinium-enhancing lesions on a single MRI scan
   * ≥1 T1 gadolinium-enhancing lesions on two or more separate MRI scans
   * ≥2 new T2 lesions compared to a previous scan within a period ≤1 year

     * Ambulatory patients (EDSS of 3 to 6 points, inclusive assessed outside of relapse)
     * Disease duration less than 15 years
     * Participants must receive or be current on all recommended vaccinations according to institutional, local, or global guidelines for immunocompromised patients at least 6-weeks prior to lymphodepletion

Exclusion Criteria:

* Diagnosis of primary progressive multiple sclerosis (PPMS) according to the 2017 revision of the McDonald diagnostic criteria at screening
* History of or current clinically significant CNS disease (e.g. stroke, traumatic brain or spinal injury, history or presence of myelopathy) or neurological disorders which may mimic MS or ICANS at screening
* Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 6 months prior to screening), neurological disorders other than MS (including seizure disorders even when well controlled), psychiatric, pulmonary (including, history of or active severe respiratory disease, including Chronic Obstructive Pulmonary Disease, interstitial lung disease or pulmonary fibrosis), renal, hepatic, endocrine, metabolic (e.g. severe hypoproteinemia due to nephrotic syndrome), hematological disorders or gastrointestinal disease that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant, prior to screening
* Have donated blood or experienced a loss of blood > 400 mL within 3 months prior screening, or longer if required by local regulations
* Any prior stem cell therapy or organ transplantation or gene therapy
* Any contraindications to LP, including but not limited to:

  * Known or suspected structural abnormality of the lumbar spine that, in the opinion of the Investigator, may interfere with the performance of the LP, or increase the risk of the procedure for the participant
  * Presence of risk for increased or uncontrolled bleeding including, but not limited to, vascular abnormalities or neoplasms at or near the LP site, disorders of the coagulation cascade, platelet function, or platelet count
  * Participants on anticoagulants (e.g., warfarin) or antiplatelets [except for low-dose aspirin (100 mg/day or lower) and low-dose ibuprofen (600 mg/day or lower) which are allowable], are not eligible to participate
* Participants not willing or able to take MRI scans as per protocol. Unable to undergo MRI due to for example claustrophobia, or presents absolute contraindications to MRI (e.g., metallic implants, metallic foreign bodies, pacemaker, defibrillator)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 through Year 2
  Incidence of dose limiting toxicities (DLTs), AEs and SAEs, including changes in vital signs, electrocardiograms (ECGs), laboratory parameters, neurological status and magnetic resonance (MRI) of the brain and spinal cord qualifying and reported as AEs.

SECONDARY OUTCOMES:
Measure of Disability: Expanded Disability Status Scale (EDSS). | Day 1 through Year 2
  EDSS is used to measure the change in disability level in participants using a scale from 0 to 10. The higher the score, the greater the degree of disability.
Measure of Disability: Short Form Health Survey (SF-36 v2) | Day 1 through Year 2
  The Short Form Health Survey (SF-36 v2) is a widely used and extensively studied instrument to measure health-related quality of life among healthy participants and participants with acute and chronic conditions. It consists of eight subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) also can be computed. The SF 36 has proven useful in monitoring general and specific populations, comparing the relative burden of different diseases, differentiating the health benefits produced by different treatments, and in screening individual participants.
Measure of Disability: Timed 25 Foot Walk (T25FW) | Day 1 through Year 2
  The T25FW is a mobility test based on a timed walk of 25 feet that is administered by a trained administrator. The participant is directed to walk the clearly marked 25-foot distance as quickly as possible. Longer completion time corresponds with decreased mobility.
Measure of Disability: 9 Hole Peg Test (9HPT) | Day 1 through Year 2
  The 9HPT is a finger dexterity test that is administered by a trained administrator. The participant is directed to put 9 pegs, one by one, onto and then off the holder board as quickly as possible starting with using only the dominant hand, and then repeated with the non-dominant hand. Longer completion times are associated with decreased finger dexterity.
Measure of Disability: Symbol Digit Modalities Test (SDMT) | Day 1 through Year 2
  The SDMT is a timed cognition test administered by a trained administrator. The test assesses sustained attention, processing speed, visual scanning, and motor speed to determine cognitive impairment. Participants are given a coding key which contains abstract symbols that correspond to specific numbers. Participants are timed how quickly and accurately they are able to substitute the symbols for the numbers and is scored by the number of correctly coded items.
Measure of Disability: Fatigue Symptoms and Impacts Questionnaire - Relapsing Multiple Sclerosis (FSIQ-RMS) | Day 1 through Year 2
  The FSIQ-RMS is a questionnaire to assess fatigue-related symptoms in patients with RMS. Participants will indicate the severity of fatigue experienced for each question that examines different aspects of fatigue.
Number of new and enlarging T2 lesions and Gd-enhancing T1 Lesions | Day 1 through Year 2
  Measured in the brain by Magnetic Residence Imaging (MRI)
Plasma Pharmacokinetics (PK) of YTB323 - CMAX | Day 1 through Year 2
  Measured by Cmax - The maximum plasma concentration of YTB323
Plasma Pharmacokinetics (PK) of YTB323 - AUC | Day 1 through Year 2
  Measured by AUC - Area under the curve of YTB323
Plasma Pharmacokinetics (PK) of YTB323 - Tmax | Day 1 through Year 2
  Measured by Tmax - Time to Reach the Maximum Concentration After Drug Administration of YTB323
Plasma Pharmacokinetics (PK) of YTB323 - Clast | Day 1 through Year 2
  Clast is defined as the Last observed (quantifiable) plasma concentration (Clast)
Plasma Pharmacokinetics (PK) of YTB323 - Tlast | Day 1 through Year 2
  Tlast is defined as Time of Last Measurable Concentration
Safety data including dose limiting toxicities (DLTs), Adverse Events (AEs), and Serious Adverse Events (SAEs) from each dose level | Day 1 through Year 2
  Safety data from each dose level will be used to assess safe dose-level(s) to be continued in phase 2 and later clinical studies
Humoral Immunogenicity of YTB323 | Day 1 through Year 2
  Incidence and prevalence of pre-existing and treatment induced humoral immunogenicity of YTB323
Cellular Immunogenicity of YTB323 | Day 1 through Year 2
  Incidence and prevalence of pre-existing and treatment induced cellular immunogenicity of YTB323

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- France (3):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Rennes
- Germany (3):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Ulm
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
- Spain (4):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com